CLINICAL TRIAL: NCT01483495
Title: Assessing Cerebrovascular Reactivity Based on Cerebral Oximetry
Brief Title: Assessing Cerebrovascular Reactivity Based on Cerebral Oximetry: a Pilot Study
Acronym: DOSI
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Lingzhong Meng, M.D.,Assistant Clinical Professor and Director of Neuroanesthesia, University of California, Irvine
Other Study IDs: 20107521
Record Dates: First submitted 2011-08-02; First posted 2011-12-01 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Hypoxia-Ischemia, Brain; Signs and Symptoms
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Signs and Symptoms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnostic tool: Diffuse Optical Spectroscopy Imaging Cerebrovascular Reactivity
  Interventions: Device: Diffuse optical spectroscopy

INTERVENTIONS:
Device: Diffuse optical spectroscopy — Diffuse Optical Spectroscopy Imaging Cerebrovascular Reactivity
  Other Names: Diffuse Optical Spectroscopy Imaging

SUMMARY:
The brain is such a metabolically active organ that it consumes about 20% of oxygen burned every minute by an average adult even though it only contributes about 2% of the body weight. As a result, the brain produces a disproportionately high amount of CO2 every minute in comparison with the rest of the body.

DETAILED DESCRIPTION:
The researcher can use Diffuse Optical Spectroscopy Imaging, cerebral non-invasive oximetry instrument, to determine cerebrovascular reactivity during surgery procedure. Specifically, the cerebral tissue O2 saturation can measure by Diffuse Optical Spectroscopy Imaging can use for cerebral blood flow in the evaluation of cerebrovascular reactivity.

Adequate brain perfusion is critical not only to supply oxygen and nutrients but also to wash out metabolic end products including CO2. Blood flow depends on perfusion pressure and vascular bed resistance. It is well known that multiple physiological and pathological factors affect cerebral vasculature, and the resistance to blood flow. The cerebrovascular responsiveness to those factors determines how well the brain can maintain and adjust its perfusion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female 20 years of age and older
2. Female non-pregnant
3. Subject scheduled for elective surgery under general anesthesia with intubation.
4. Subject who is able to give informed consent.

Exclusion Criteria:

1. Less than 20 years old of age
2. Pregnant woman
3. Subjects currently diagnosed with severe hypertension, myocardial ischemic disease, symptomatic valvular disease(s), symptomatic arrhythmia, uncompensated congestive heart failure, intracranial aneurysm.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2011-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Brain blood flow | 6 hours
  Optical Imaging assess of Brain blood flow during surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Tromberg, PhD, Study Director — Beckman Laser Institute; Lingzhong Meng, M.D, Principal Investigator — Anesthesiology Perioperative Care
Locations (1):
- UCI Beckman Laser Institute, Irvine, California, United States